CLINICAL TRIAL: NCT05602597
Title: A Phase 1, Open-Label, 4-Part, Fixed-Sequence Study to Assess the Effect of Itraconazole, a Strong CYP3A Inhibitor, the Effect of Fluconazole, a Moderate CYP3A/2C9 Inhibitor, the Effect of Rifampin, a Strong CYP3A Inducer, and the Effect of Rabeprazole, a Proton Pump Inhibitor on the Pharmacokinetics of HMPL-689 in Healthy Volunteers
Brief Title: HMPL-689 Drug Interaction Study With CYP3A Inhibitor/CYP2C9 Inhibitor/CYP3A Inducer/PPI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2021-689-00US1
Record Dates: First submitted 2022-10-27; First posted 2022-11-02 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Relapsed or Refractory Lymphoma
Keywords: Itraconazole; Fluconazole; Rifampin; Rabeprazole
MeSH Terms: conditions — Recurrence; Lymphoma | interventions — Itraconazole; Fluconazole; Rifampin; Rabeprazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A - Itraconazole (Experimental): Period 1 -- Participants to receive 10mg dose of HMPL-689 by mouth as a single agent treatment on Day 1
  Period 2 -- Participants to receive 200mg Itraconazole by mouth twice daily beginning on Day 3 through Day 10. On Day 7 200 mg Itraconazole and 10 mg HMPL-689 will be simultaneously administered.
  Interventions: Drug: Itraconazole 200 mg
- Part B - Fluconazole (Experimental): Period 1 -- Participants to receive 10mg dose of HMPL-689 by mouth as a single agent treatment on Day 1
  Period 2 -- Participants to receive 400mg Fluconazole by mouth daily on Day 3, then 200 mg Fluconazole by mouth daily Day 4 through Day 10. On Day 7 200 mg Fluconazole and 10 mg HMPL-689 will be simultaneously administered.
  Interventions: Drug: Fluconazole 400 mg
- Part C - Rimfampin (Experimental): Period 1 -- Participants to receive 30mg dose of HMPL-689 by mouth as a single agent treatment on Day 1
  Period 2 -- Participants to receive 600mg Rifampin by mouth daily beginning on Day 3 through Day 11. On Day 10 600mg Rifampin will be administered by mouth approximately 1 hour before the start of breakfast and 30mg HMPL-689 will be administered by mouth approximately 30 minutes after the start of breakfast.
  Interventions: Drug: Rifampin 600 mg
- Part D - Rabeprazole (Experimental): Period 1 -- Participants to receive 30mg dose of HMPL-689 by mouth as a single agent treatment on Day 1
  Period 2 -- Participants to receive 40mg Rabeprazole by mouth daily beginning on Day 3 through Day 9. On Day 9 40mb Rabeprazole will be administered by mouth approximately 1 hour before the start of breakfast and 30mg HMPL-689 will be administered by mouth approximately 30 minutes after the start of breakfast.
  Interventions: Drug: Rabeprazole 40 mg

INTERVENTIONS:
Drug: Itraconazole 200 mg — Study participants will be administered 200 mg itraconazole by mouth twice daily after the pharmacokinetic blood draw on Day 3 and once daily on Days 4 to 10, inclusive.
  Arms: Part A - Itraconazole
Drug: Fluconazole 400 mg — Study participants will be administered 400 mg fluconazole by mouth daily on Day 3 after the pharmacokinetic blood draw, and 200 mg fluconazole by mouth daily on Days 4 to 10, inclusive.
  Arms: Part B - Fluconazole
Drug: Rifampin 600 mg — Study participants will be administered 600 mg rifampin by mouth daily starting on Day 3, after the pharmacokinetic blood draw, and on Days 4 to 11, inclusive.
  Arms: Part C - Rimfampin
Drug: Rabeprazole 40 mg — Study participants will be administered 40 mg rabeprazole by mouth daily on Day 3, after the pharmacokinetic blood draw, and on Days 4 to 9, inclusive.
  Arms: Part D - Rabeprazole

SUMMARY:
An open-label study to determine effect of Itraconazole, Fluconazole, Rifampin, and Rabeprazole on the PK of HMPL-689

DETAILED DESCRIPTION:
A phase 1, open-label, 4-part, 2-period, fixed-sequence study to assess the effect of Itraconazole, a strong CYP3A inhibitor, the effect of Fluconazole, a moderate CYP3A/2C9 inhibitor, the effect of Rifampin, a strong CYP3A inducer, and the effect of Rabeprazole, a proton pump inhibitor on the pharmacokinetics (PK) of a single oral dose of HMPL-689 in study participants. The secondary objective is to evaluate the safety of a single oral dose of HMPL-689 administered with and without Itraconazole, Fluconazole, Rifampin, or Rabeprazole in study participants.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female between the ages of 18 and 55 years old (inclusive) at the time of informed consent.
2. Body mass index (BMI) >18 and ≤29.9 kg/m2 at screening.
3. Females must be postmenopausal (defined as absence of menses for at least 1 year without alternative medical cause) or permanently sterile by total hysterectomy, bilateral oophorectomy, or bilateral salphingectomy.
4. Males, including those who have had a successful vasectomy, must use a condom during sexual intercourse with women of childbearing potential starting from their first dose of study drug through 30 days after their last dose of study drug. Alternatively, abstinence is allowed if it is the normal and preferred lifestyle of the healthy volunteer.
5. Must provide written informed consent prior to any study-specific screening procedures.
6. Willing and able to comply with all aspects of the protocol, as determined by the PI.

Exclusion Criteria:

1. Known history of any gastrointestinal surgery or any condition possibly affecting drug absorption (eg, cholecystectomy, gastrectomy, achlorhydria, peptic ulcer disease, history of stomach or intestinal surgery, or resection). Appendectomy and hernia repair are allowed.
2. Clinically significant illness within 8 weeks or a clinically significant infection within 4 weeks prior to the first dose.
3. Evidence of a clinically significant deviation from normal in the physical examination, vital signs, or clinical laboratory determinations at screening or at Day -1 Check-in (baseline).
4. Systolic blood of pressure >140 mmHg or diastolic blood pressure of > 90 mmHg.
5. Clinically significant ECG abnormality, including a marked baseline prolongation of QT/QTc interval (eg, repeated demonstration of a QTcF interval of > 450 msec), or had a family history of prolonged QTc syndrome or sudden death.
6. History of smoking or use of nicotine containing substances within the previous 2 months, as determined by medical history or healthy volunteer's verbal report and confirmed by cotinine test at check in for each treatment period.
7. History of drug and/or alcohol misuse prior to screening or a positive urine drug test at Screening or at Check in for each treatment period.
8. Diagnosed with acquired immune deficiency syndrome or has performed tests that are positive for human immunodeficiency virus, hepatitis B virus (HBV), hepatitis C virus (HCV), cytomegalovirus, or pneumocystis jiroveci pneumonia.
9. Participated in a clinical trial of other drug before screening, and the time since the last use of other study drug is less than 5 times the half-life or 4 weeks, whichever is longer, or the healthy volunteer is currently enrolled in another clinical study.
10. Consumed grapefruit, starfruit, Seville oranges, or their products within 7 days prior to the first dose.
11. Consumed herbal preparations/medications, including, but not limited to, St. John's Wort, kava, ephedra (ma huang), Ginkgo biloba, dehydroepiandrosterone, yohimbe, saw palmetto, and ginseng, within 7 days prior to the first dose (21 days for St. John's Wort).
12. Experienced a weight loss or gain of >10% within 4 weeks prior to the first dose as noted by medical history and weight at screening and Check-in.
13. Received blood or blood products within 4 weeks or donated blood or blood products within 8 weeks prior to the first dose or donated double red cell within 16 weeks prior to first dose.
14. Used any over-the-counter (OTC) medications or prescription drugs (medications that can inhibit or induce CYP3A4/CYPC9, or lower gastric acid in particular) within 2 weeks prior to the first dose.
15. Allergic to any of the study drugs (or its excipients) to be given in this study.
16. Female healthy volunteer is pregnant, lactating, or breastfeeding.
17. Male healthy volunteer who plans to donate sperm or father a child within 30 days after receiving the study drug.
18. Any condition that would make him or her, in the opinion of the PI or sponsor, unsuitable for the study, or who, in the opinion of the PI, is not likely to complete the study for any reason.
19. For Part A only, participants characterized by any of the following CYP2C9 genotypes: *2/*2, *2/*3, or *3/*3.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-08-06 (Actual); Study Completion 2022-08-06 (Actual)

PRIMARY OUTCOMES:
AUC0-t | From Day 1 to Day 11 (Day 12 for Rifampin)
  Area under the plasma concentration-time curve from time 0 to time of the last measurable concentration
AUC0-inf | From Day 1 to Day 11 (Day 12 for Rifampin)
  Area under the plasma concentration-time curve from time 0 to infinity (if data permit)
Cmax | From Day 1 to Day 11 (Day 12 for Rifampin)
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Incidence of AEs/SAEs | From Day 1 to Day 11 (Day 12 for Rifampin)
  Any untoward medical occurrence associated with the use of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Jayaprakash, MD, Study Director — Hutchmed
Locations (1):
- QPS- Miami, Miami, Florida, United States